CLINICAL TRIAL: NCT07340216
Title: An Open Label, Phase 1, Maximal Usage Pharmacokinetics and Safety Study of ARQ-154 Foam 0.3% Administered QD in Pediatric Participants With Scalp and Body Psoriasis
Brief Title: Maximal Usage Pharmacokinetics and Safety Study of ARQ-154 Foam 0.3% in Pediatric Participants With Scalp and Body Psoriasis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ-154-127
Record Dates: First submitted 2025-12-19; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Psoriasis
Keywords: Scalp and Body Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARQ-154 Foam 0.3% (Experimental): ARQ-154 foam 0.3% will be applied QD. Treatment duration will be up to 6 weeks, including 2 weeks under maximal usage conditions, followed by an optional 4 weeks under non-maximal usage conditions.
  Interventions: Drug: ARQ-154 Foam 0.3%

INTERVENTIONS:
Drug: ARQ-154 Foam 0.3% — ARQ-154 Foam 0.3%

SUMMARY:
This study will evaluate the systemic exposure and characterize the plasma pharmacokinetic (PK) profile and assess the safety and tolerability of ARQ-154 foam 0.3%.

DETAILED DESCRIPTION:
ARQ-154-127 is a Phase 1, open-label, single arm, maximum usage pharmacokinetic and safety study of roflumilast foam 0.3% in participants with scalp and body psoriasis.

The goal of the study is to:

* Evaluate the systemic exposure and characterize the plasma pharmacokinetic (PK) profile of ARQ-154 foam 0.3%.
* Assess the safety and tolerability of ARQ-154 foam 0.3%

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 2 years to < 12 years old at Day 1.
* Clinical diagnosis of psoriasis vulgaris of at least 2 months duration at Screening as determined by the Investigator.
* Scalp psoriasis with an Investigator Global Assessment (S-IGA) of scalp disease severity of at least Moderate ('3') at Day 1.
* An IGA of body (non-scalp) psoriasis (B-IGA) of at least Mild ('2') at Day 1.
* Extent of scalp psoriasis involving ≥ 10% of the total scalp at Day 1.
* Body psoriasis (non-scalp) involving at least 3% BSA on Day 1.

Exclusion Criteria:

* Participants who cannot discontinue medications and treatments prior to Day 1 (first application of IP).
* Current diagnosis of non-plaque forms of psoriasis. Current diagnosis of drug-induced psoriasis.
* Participants who have significant active systemic or localized infection or have had any infection that required oral or intravenous administration of antibiotics, antifungal or antiviral agents within 7 days prior to Day 1.
* Participants with skin conditions other than psoriasis vulgaris that would interfere with evaluations of the effect of the study medication, as determined by the Investigator.
* Participants who cannot discontinue the use of strong cytochrome P-450 CYP3A4 inhibitors for 2 weeks prior to Day 1 and during the study period.
* A medical history of severe renal insufficiency, moderate to severe hepatic disorders (e.g., Child-Pugh B or C), or chronic infectious disease (e.g., hepatitis B, hepatitis C, or human immunodeficiency virus [HIV]).
* Participants who are family members of the clinical study staff or sponsor.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Concentration of Roflumilast and Roflumilast N-Oxide from plasma | 2 Weeks
  Assessment of steady-state trough plasma concentrations after 2 weeks of study drug administration.
Participant incidence of adverse events | 6 Weeks
  Number of participants with adverse events during treatment will be assessed
Incidence of application site reactions | 6 Weeks
  Number of participants that experience an application site skin reaction by investigator assessment and participant assessment will be assessed
The incidence of changes from Baseline in the total Children's Depression Inventory 2 (CDI-2)score. | 6 Weeks
  The CDI-2 is an assessment instrument used to evaluate the severity of depressive symptoms in children.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Arcutis Clinical Study Site 106, Bryant, Arkansas
  - Arcutis Clinical Study Site 107, Miami Lakes, Florida
  - Arcutis Clinical Study Site 108, Meridian, Idaho
  - Arcutis Clinical Study Site 105, West Lafayette, Indiana
  - Arcutis Clinical Study Site 104, Arlington, Texas